CLINICAL TRIAL: NCT02864043
Title: Identification of Features Associated With Dysplasia Using the NvisionVLE® Imaging System Pilot Trial
Brief Title: Barrett's Dysplasia Detection Pilot Trial Using the NvisionVLE® Imaging System
Acronym: DDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-01
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Barrett's; OCT; VLE
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EGD with NvisionVLE with Real Time Targeting (Other): Physician will complete a VLE scan of the esophagus and target areas of interest using the VLE optical marking probe following standard of care endoscopy
  Interventions: Device: NvisionVLE with Real Time Targeting; Procedure: esophagogastroduodenoscopy (EGD)

INTERVENTIONS:
Device: NvisionVLE with Real Time Targeting — Physician will complete a VLE scan of the esophagus and target areas of interest using the VLE optical marking probe
Procedure: esophagogastroduodenoscopy (EGD) — Standard of care EGD

SUMMARY:
The NvisionVLE® Dysplasia Detection Pilot Study is a prospective, non-randomized trial for participants who have a prior biopsy-confirmed diagnosis of BE with dysplasia and are scheduled to have an endoscopic evaluation of your esophagus for BE surveillance by a standard procedure called EGD (esophagogastroduodenoscopy) as well as an imaging procedure called VLE (volumetric laser endomicroscopy).

DETAILED DESCRIPTION:
The NvisionVLE® Dysplasia Detection Pilot Study is a collection of data for research. Participation is completely voluntary and does not affect the patient's medical care that chooses not to participate. The purpose of this Study is to determine the performance of the NvisionVLE® Imaging System in determining features of dysplastic Barrett's Esophagus (BE). This is done by the collection and analysis of the medical record information, imaging data, and pathology results. The information is then stored and may be used at a later time for various future analyses and publications. Any future analyses involving this Study will only use the information collected in this Study. No further involvement or additional informed consent of participants will be needed if future analyses are performed.

This Study is designed for participants who have a prior biopsy-confirmed diagnosis of BE with dysplasia and are scheduled to have an endoscopic evaluation of your esophagus for BE surveillance by a standard procedure called EGD (esophagogastroduodenoscopy) as well as an imaging procedure called VLE (volumetric laser endomicroscopy).

The NvisionVLE® Imaging System is cleared for use by the U.S. Food and Drug Administration (FDA).

Patients who undergo an endoscopic evaluation of the esophagus with the NvisionVLE® Imaging System at participating hospitals will be invited to participate in this Study. The Study is taking place at up to 4 hospitals, and as many as 100 patients may participate in this Study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18.
* Patients undergoing an upper endoscopy for BE surveillance with prior biopsy-confirmed BE with dysplasia (at least LGD).
* Ability to provide written, informed consent.
* No significant esophagitis (LA grade < B, C and D).

Exclusion Criteria:

* Patients who have achieved complete remission of intestinal metaplasia (CR-IM)
* Patients without visible BE at time of study EGD.
* Patients for whom use of the NvisionVLE device would be in conflict with the Instructions for Use (IFU).
* Prior esophageal or gastric surgical resection.
* Significant esophageal stricture requiring dilatation.
* Patients who require anticoagulation for whom biopsy would be contraindicated.
* Patients who are known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Performance of manually identified VLE features in predicting biopsy defined dysplasia | Up to 2 years post data collection
  To determine the per-biopsy performance of a multivariable model consisting of manually-identified VLE features for predicting biopsy-defined dysplasia

SECONDARY OUTCOMES:
Per Patient Sensitivity and specificity for detecting dysplasia | Up to 2 years post data collection
  1. To determine the absolute per-patient sensitivity and specificity of a multivariable model consisting of manually-identified VLE features for predicting biopsy-defined dysplasia.
Per Biopsy Sensitivity and specificity for detecting dysplasia | Up to 2 years post data collection
  2. To determine the absolute per-biopsy sensitivity and specificity of a multivariable model consisting of manually-identified VLE features for predicting biopsy-defined dysplasia.
Per Biopsy performance of VLE compared to standard-of-care for detecting dysplasia | Up to 2 years post data collection
  3. To compare, on a per-biopsy basis, the performance of VLE and standard-of-care to standard-of-care alone in detecting dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wang, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - UC Irvine Medical Center, Irvine, California
  - VA Boston, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No